CLINICAL TRIAL: NCT01896895
Title: Prospective, Double-blind, Placebo-controlled, Randomized, Parallel-group, Multi-center Study With an Open-label Extension Period to Investigate the Efficacy and Safety of Two Different Doses of NT 201 in Botulinum Toxin Treatment-naïve Subjects With Blepharospasm
Brief Title: Efficacy and Safety Study of Botulinum Toxin Type A Against Placebo to Treat Abnormal Contraction or Twitch of the Eyelid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Pharmaceuticals GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MRZ60201_3074_1; 2012-004821-26 (EudraCT Number)
Record Dates: First submitted 2013-07-08; First posted 2013-07-11 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-01

CONDITIONS: Bilateral Blepharospasm (BEB)
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- IncobotulinumtoxinA (Xeomin) 25U per eye (Experimental): Main Period: one injection session, 25 Units per eye. Open-Label Extension: one injection session, up to 35 Units per eye. Mode of administration: intramuscular injection.
  Interventions: Drug: IncobulinumtoxinA (Xeomin), 25 Units; Drug: IncobotulinumtoxinA (Xeomin), 35 Units
- IncobotulinumtoxinA (Xeomin) 12.5U per eye (Experimental): Main Period: one injection session, 12.5 Units per eye. Open-Label Extension Period: one injection session, up to 35 Units per eye. Mode of administration: intramuscular injection.
  Interventions: Drug: IncobotulinumtoxinA (Xeomin), 12.5 Units; Drug: IncobotulinumtoxinA (Xeomin), 35 Units
- Placebo (Placebo Comparator): Main Period: Placebo to IncobotulinumtoxinA (Xeomin)(12.5 or 25U/eye), one injection session.
  Open-Label Extension: IncobotulinumtoxinA (Xeomin), one injection session, up to 35 Units per eye. Mode of administration: intramuscular injection.
  Interventions: Drug: Placebo; Drug: IncobotulinumtoxinA (Xeomin), 35 Units

INTERVENTIONS:
Drug: IncobulinumtoxinA (Xeomin), 25 Units — IncobotulinumtoxinA (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl). Main Period: 25 Units per eye.
  Other Names: NT 201; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: IncobotulinumtoxinA (Xeomin) 25U per eye
Drug: IncobotulinumtoxinA (Xeomin), 12.5 Units — IncobotulinumtoxinA (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl). Main Period: 12.5 Units per eye.
  Other Names: NT 201; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
  Arms: IncobotulinumtoxinA (Xeomin) 12.5U per eye
Drug: Placebo — Main Period: Placebo to IncobotulinumtoxinA (Xeomin), powder for solution for injection, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Arms: Placebo
Drug: IncobotulinumtoxinA (Xeomin), 35 Units — IncobotulinumtoxinA (active ingredient: Clostridium Botulinum neurotoxin Type A free from complexing proteins) powder for solution for injection, prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl).
  Open-Label Extension: up to 35 Units per eye.
  Other Names: NT 201; Xeomin; Botulinum toxin type A (150 kiloDalton), free from complexing proteins

SUMMARY:
This phase 3 study will serve to collect efficacy and safety data of two different doses of NT 201 in subjects suffering from Bilateral Blepharospasm (BEB) who are BTX treatment-naïve.

In this study, BTX treatment-naïve subjects are defined as those who have not received BTX treatment within the last 12 months for the treatment of BEB. This definition aims to avoid bias by comparison of treatment effects in the subject's assessments. Furthermore, this study will substantiate the existing efficacy and safety database for the indication BEB.

DETAILED DESCRIPTION:
Subjects to receive one injection with NT 201 or placebo at baseline of the placebo-controlled first cycle. Thereafter, all subjects entering the Open-Label Extension Period (OLEX) to receive a second injection of NT 201 (second injection cycle).

ELIGIBILITY:
Inclusion Criteria:

* Male or female out-patients age ≥ 18 and ≤ 80 years.
* A clinical diagnosis of bilateral BEB characterized by spontaneous, spasmodic, intermittent or persistent involuntary contractions of orbicular oculi muscles.
* A need for injection of BTX defined as a Jankovic Rating Scale [JRS] severity subscore ≥ 2.
* Treatment-naïve subject defined as at least 12 months without BTX of any serotype for the treatment of BEB before administration of IP.

Exclusion Criteria:

* Subject with any previous unsuccessful treatment with BTX of any serotype for the treatment of BEB.
* Atypical variant of BEB (e.g., apraxia of the eyelid opening) caused by inhibition of levator palpebrae muscle.
* Neuroleptic-induced blepharospasm.
* Myotomy or denervation surgery in the affected muscles (e.g., peripheral denervation, spinal cord stimulation) and surgery in the upper face.
* Generalized disorders of muscles activity (e.g., myasthenia gravis in particular ocularis, Lambert-Eaton-Syndrome, amyotrophic lateral sclerosis) or any other significant neuromuscular dysfunction which might interfere with the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-11; Primary Completion 2016-04 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Pharmaceuticals GmbH
Locations (11):
- Greece (2):
  - Merz Investigational Site #030002, Athens
  - Merz Investigational Site #030001, Athens
- Malaysia (5):
  - Merz Investigational Site #060007, George Town, Pulau Pinang
  - Merz Investigational Site #060004, Kota Kinabalu, Sabah
  - Merz Investigational Site #060006, Kuala Lumpur
  - Merz Investigational Site #060002, Kuala Lumpur
  - Merz Investigational Site #060003, Kuala Selangor
- Sri Lanka (4):
  - Merz Investigational Site #094001, Colombo
  - Merz Investigational Site #094005, Colombo
  - Merz Investigational Site #094006, Kurunegala
  - Merz Investigational Site #094002, Nugegoda

REFERENCES:
- [Derived] Mitsikostas DD, Dekundy A, Hanschmann A, Althaus M, Scheschonka A, Pagan F, Jankovic J. Duration and onset of effect of incobotulinumtoxinA for the treatment of blepharospasm in botulinum toxin-naive subjects. Curr Med Res Opin. 2021 Oct;37(10):1761-1768. doi: 10.1080/03007995.2021.1965975. Epub 2021 Aug 24. PMID 34384301
- [Derived] Duarte GS, Rodrigues FB, Marques RE, Castelao M, Ferreira J, Sampaio C, Moore AP, Costa J. Botulinum toxin type A therapy for blepharospasm. Cochrane Database Syst Rev. 2020 Nov 19;11(11):CD004900. doi: 10.1002/14651858.CD004900.pub3. PMID 33211907
- [Derived] Mitsikostas DD, Dekundy A, Sternberg K, Althaus M, Pagan F. IncobotulinumtoxinA for the Treatment of Blepharospasm in Toxin-Naive Subjects: A Multi-Center, Double-Blind, Randomized, Placebo-Controlled Trial. Adv Ther. 2020 Oct;37(10):4249-4265. doi: 10.1007/s12325-020-01427-6. Epub 2020 Aug 10. PMID 32779096

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 68 participants were screened, 61 were enrolled and treated of which 55 completed the double-blind main period (MP). 39 participants from the double-blind MP entered the Open label Extension (OLEX) period and completed the study.
Groups:
- Double-blind MP: Placebo: Participants received 1.0 milliliter (mL) placebo matched to the volume of incobotulinumtoxinA doses per injection session via intramuscular injections into orbicular oculi muscles on Day 1 in the double-blind MP.
- Double-blind MP: IncobotulinumtoxinA 25 Units: Participants received 1.0 mL of incobotulinumtoxinA containing 25 units per injection session (12.5 units per eye) via intramuscular injections into orbicular oculi muscles on Day 1 in the double-blind MP.
- Double-blind MP: IncobotulinumtoxinA 50 Units: Participants received 1.0 mL of incobotulinumtoxinA containing 50 units per injection session (25 units per eye) via intramuscular injections into orbicular oculi muscles on Day 1 in the double-blind MP.
- OLEX: IncobotulinumtoxinA 70 Units: Participants received up to 1.4 mL of incobotulinumtoxinA containing up to 70 units per injection session (35 units per eye) via intramuscular injections into orbicular oculi muscles on Day 1 in the OLEX Period.
Period: Double-blind MP
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units | OLEX: IncobotulinumtoxinA 70 Units
Started | 20 | 22 | 19 | 0
Completed | 19 | 20 | 16 | 0
Not Completed | 1 | 2 | 3 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0
Period: OLEX Period
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units | OLEX: IncobotulinumtoxinA 70 Units
Started | 0 | 0 | 0 | 39 (Not all participants who completed double-blind MP fulfilled the inclusion criteria for OLEX period.)
Completed | 0 | 0 | 0 | 39
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) was subset of participants in the safety evaluation set (SES) of the double-blind MP for whom at least a baseline value of the Jankovic Rating Scale (JRS) severity subscore was available.
Groups:
- Double-blind MP: Placebo: Participants received 1.0 mL placebo matched to the volume of incobotulinumtoxinA doses per injection session via intramuscular injections into orbicular oculi muscles on Day 1 in the double-blind MP.
- Total: Total of all reporting groups
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units | Total
Number analyzed (Participants) | 20 | 22 | 19 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 14 | 44
  >=65 years | 3 | 9 | 5 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.4 (12.01) | 55.8 (15.70) | 53.5 (13.82) | 55.0 (13.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 11 | 13 | 36
  Male | 8 | 11 | 6 | 25
Region of Enrollment [Number; unit: participants]
  Greece | 4 | 6 | 4 | 14
  Sri Lanka | 10 | 10 | 10 | 30
  Malaysia | 6 | 6 | 5 | 17

OUTCOME MEASURES:

1. Primary Outcome: Double-blind MP: Change From Baseline in JRS Severity Subscore at Day 43 (Visit 4)
Description: JRS severity subscore was used to classify individual symptoms of blepharospasm and to determine therapeutic efficacy. JRS severity subscore ranges from 0 to 4, where 0: None; 1: increased blinking present with external stimuli; 2: Mild but spontaneous eyelid fluttering, definitely noticeable, possibly embarrassing, but not functionally disabling, 3: Moderate, very noticeable spasm of eyelids only, mildly incapacitating, 4: Severe, incapacitating spasm of eyelids and possibly other facial muscles. Values represent least square (LS) mean differences between baseline and visit 4 resulting from analysis of covariance (ANCOVA) with treatment group, pooled site, and gender as fixed factors and baseline JRS severity subscore and age as covariates and missings replaced using the last observation carried forward (LOCF) method. Negative values denote improvement, while positive values denote deterioration vs. baseline.
Time Frame: Baseline, Day 43 (Visit 4)
Population: FAS was subset of participants in the SES of the double-blind MP for whom at least a baseline value of the JRS severity subscore was available.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units
Number analyzed (Participants) | 20 | 22 | 19
score on a scale | -0.6 [-1.0 to -0.1] | -1.0 [-1.5 to -0.6] | -1.8 [-2.3 to -1.3]
Statistical Analysis 1: Comparison: Double-blind MP: Placebo vs Double-blind MP: IncobotulinumtoxinA 50 Units; The difference in change of JRS severity subscore between treatment groups was analyzed by an ANCOVA according to a hierarchical test procedure. First step of hierarchy is hypothesis of superiority of 50 unit dose group NT 201 compared to placebo. This was tested confirmatory (α=0.05, 2-sided) by an ANCOVA with treatment group, pooled site, and gender as fixed factors and baseline JRS severity subscore and age as covariates based on LS means comparison. Missing values were imputed by LOCF; Test type: Superiority; p = 0.0004, ANCOVA; LS mean difference = -1.2, 95% CI 2-sided [-1.9 to -0.6]
Statistical Analysis 2: Comparison: Double-blind MP: Placebo vs Double-blind MP: IncobotulinumtoxinA 25 Units; The difference in change of JRS severity subscore between treatment groups was analyzed by an ANCOVA according to a hierarchical test procedure. Second step of hierarchy is hypothesis of superiority of 25 unit dose group NT 201 compared to placebo. This was tested confirmatory (α=0.05, 2-sided) by an ANCOVA with treatment group, pooled site, and gender as fixed factors and baseline JRS severity subscore and age as covariates based on LS means comparison. Missing values were imputed by LOCF; Test type: Superiority; p = 0.1452, ANCOVA; LS mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.2]

2. Secondary Outcome: Double-blind MP: Change From Baseline in Blepharospasm Disability Index (BSDI) at Day 43 (Visit 4)
Description: BSDI is a scale for assessment of impairment of specific activities of daily living caused by blepharospasm. BSDI consists of six items (driving a vehicle; reading; watching TV; shopping; getting about on foot (walking); doing everyday activities), each ranging from 0 (=no impairment) to 4 (=no longer possible due to illness). The BSDI total score is a mean score for non-missing items ranging from 0 to 4. It is calculated by adding scores of all applicable and answered items, and dividing the resulting sum by the number of items answered. Outcome values represent LS mean differences between baseline and visit 4 (visit 4 value minus baseline value) resulting from ANCOVA with treatment group, pooled site, gender as fixed factors and baseline BSDI total score, age as covariates. Missings were replaced by the LOCF method. Negative values denote an improvement, while positive values denote deterioration vs. baseline.
Time Frame: Baseline, Day 43 (Visit 4)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units
Number analyzed (Participants) | 20 | 22 | 19
score on a scale | -0.4 [-0.8 to 0.0] | -0.5 [-0.9 to -0.2] | -0.7 [-1.1 to -0.3]

3. Secondary Outcome: Double-blind MP: Patient Evaluation of Global Response (PEGR) at Final Visit (Day 43-Day 141)
Description: PEGR scale is a descriptive subjective 9-point response self-rating scale ranging from "complete abolishment of signs and symptoms" (value=+4) down to "very marked worsening" (value=-4). Outcome values represent least square means at visit 4 resulting from an ANCOVA with treatment group, pooled site, gender as fixed factors and age as covariates. Missing were set to a zero effect (value=0). Positive values denote an improvement, while negative values denote deterioration.
Time Frame: Baseline, Final Visit (Day 43-Day 141)
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units
Number analyzed (Participants) | 20 | 22 | 19
score on a scale | 1.3 [0.7 to 1.9] | 1.8 [1.2 to 2.4] | 2.2 [1.5 to 2.8]

ADVERSE EVENTS:
Time Frame: Double-blind MP: From the time point of first injection up to final visit (Day 43 to 141); OLEX Period: From the time point of first injection up to end of study visit (Day 43 to 141)
Description: Adverse events were collected systematically at each visit by the investigator.
Arm/Group | Double-blind MP: Placebo | Double-blind MP: IncobotulinumtoxinA 25 Units | Double-blind MP: IncobotulinumtoxinA 50 Units | OLEX: IncobotulinumtoxinA 70 Units
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22 | 0/19 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/20 | 2/22 | 1/19 | 0/39
Other Adverse Events (participants affected / at risk) | 6/20 | 7/22 | 7/19 | 4/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MP: Placebo (N=20) | Double-blind MP: IncobotulinumtoxinA 25 Units (N=22) | Double-blind MP: IncobotulinumtoxinA 50 Units (N=19) | OLEX: IncobotulinumtoxinA 70 Units (N=39)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-blind MP: Placebo (N=20) | Double-blind MP: IncobotulinumtoxinA 25 Units (N=22) | Double-blind MP: IncobotulinumtoxinA 50 Units (N=19) | OLEX: IncobotulinumtoxinA 70 Units (N=39)
Blood creatine increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid ptosis (Eye disorders) | 0 (0) | 2 (2) | 3 (3) | 2 (2)
Blepharospasm (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye pruritus (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eyelid disorder (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Periorbital oedema (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injection site erythema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.